CLINICAL TRIAL: NCT00619801
Title: A Multi-Center, Randomized, Double Blind, Placebo Controlled Parallel Group Study of the Safety of Levocetirizine Dihydrochloride Oral Liquid Formulation b.i.d Dosing in Children Aged 1 to < 6 Years Suffering From Allergic Rhinitis or Chronic Urticaria of Unknown Origin
Brief Title: Safety Study of Levocetirizine Dihydrochloride Oral Liquid Formulation in Children Aged 1 to Less Than 6 Years Suffering From Allergic Rhinitis or Chronic Urticaria of Unknown Origin
Acronym: PAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A00426; RPCE07K2404; 2015-000205-39 (EudraCT Number)
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Rhinitis; Chronic Urticaria
Keywords: Xyzal; Levocetirizine; Allergy; Children; Seasonal Allergies
MeSH Terms: conditions — Rhinitis, Allergic; Chronic Urticaria; Hypersensitivity; Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Levocetirizine (Experimental)
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — Levocetirizine dihydrochloride 1.25 mg oral drops formulation (5 drops containing 5mg/mL) dosed twice a day for 2 weeks
  Other Names: Xyzal
  Arms: Levocetirizine
Drug: Placebo — Placebo oral drops (5 drops) dosed twice a day for 2 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety of the oral formulation of levocetirizine in children ages 1 to less than 6 years old who suffer from allergic rhinitis or chronic urticaria of unknown origin.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female pediatric subject, ages 1 to less than 6 years old at the Randomization Visit (V2) (1 - < 6 years old)
* The subject must present at least one of the following symptoms, most commonly associated with allergic rhinitis or chronic urticaria: nasal itching, sneezing, rhinorrhea, nasal congestion, tearing, eye redness and itching of eyes, ears and/or palate, skin wheals and itching of the skin
* Subjects (age 2 to less than 6 years only) suffering from allergic rhinitis (AR) should have a documented allergy measured by positive skin prick test or RAST (Radioallergosorbent Test) performed within the last 6 months prior to randomization
* Candidate for antihistamine treatment or received antihistamine in the past for similar symptoms as those presenting
* Caregiver(s) have been informed of the nature and aims of the study and have given their written informed consent for the subject to participate in this study
* Caregiver(s) able to understand information given, the text of the informed consent, and be able to complete the daily record card (DRC)

Exclusion Criteria:

* Any clinically significant medical condition or abnormality other than the primary diagnosis for which an antihistamine is indicated
* Be initiating or changing the dose of an immunotherapy regimen during the course of the study (Visit 1 to Visit 4)
* Any electrocardiogram (ECG) parameters, including a QTcF interval > 443 msec measured by an ECG obtained at the Screening Visit, outside the normal reference ranges
* Any clinical laboratory tests performed at the Screening Visit, other than those related with the allergic condition, outside the reference ranges. Subjects having values outside the accepted reference range can be included if in the Investigator's opinion, they are of no clinical significance
* Personal history of seizure, febrile seizure or sleep apnea
* Below the lower 5th or above 95th percentile for body weight and/or height based upon CDC Growth Charts for Body Weight and Length
* Allergy or intolerance to levocetirizine dihydrochloride or its excipients, or to any other piperazine derivatives, such as hydroxyzine, cetirizine, cyclizine, meclozine, buclizine
* Current or past intake of the following medications (including exposure through breast milk) within the specified wash-out period before the Randomization Visit (V2):

  1. Systemic corticosteroids within the past 28 days
  2. Leukotriene-receptor antagonists (e.g. montelukast [Singulair] or zafirlukast [Accolate] within the past 7 days)
  3. Mast-cell stabilizers (e.g. cromolyn or nedocromil) within the past 7 days
  4. Other antihistamines or cough and cold preparations (with the exception of single ingredient guaifenesin products) or over-the-counter (OTC) sleep aid medications within the past 7 days
  5. Systemic antibiotics within the past 7 days
  6. Other concomitant medications that will interfere with the study, in the opinion of the investigator
* Previous participation in another clinical/pharmacological trial within the past month prior to V1
* Have already participated in this study or participated in this study at another site
* Children of any member of the study site staff

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (28):
- United States (28):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Crescent City, California
  - Huntington Beach, California
  - Mission Viejo, California
  - San Diego, California
  - Wildomar, California
  - Denver, Colorado
  - Pueblo, Colorado
  - Savannah, Georgia
  - Stockbridge, Georgia
  - Normal, Illinois
  - Overlook Park, Kansas
  - Owensboro, Kentucky
  - Metarie, Louisiana
  - Baltimore, Maryland
  - Omaha, Nebraska
  - Papillon, Nebraska
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Barnwell, South Carolina
  - Charleston, South Carolina
  - Dallas, Texas
  - El Paso, Texas
  - New Braunfels, Texas
  - Richmond, Virginia

REFERENCES:
- [Derived] Hampel F, Ratner P, Haeusler JM. Safety and tolerability of levocetirizine dihydrochloride in infants and children with allergic rhinitis or chronic urticaria. Allergy Asthma Proc. 2010 Jul-Aug;31(4):290-5. doi: 10.2500/aap.2010.31.3349. PMID 20819318
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (5 drops) dosed by mouth at breakfast time and in the evening (the evening dose should be administered approximately 12 hours later), twice a day for 2 weeks from Visit 2 (Day 0) to Visit 4 (Day 14) or the Early Discontinuation Visit (EDV).
- Levocetirizine: Levocetirizine dihydrochloride 1.25 mg (5 drops containing 5 mg/mL) dosed by mouth at breakfast time and in the evening (the evening dose should be administered approximately 12 hours later), twice a day for 2 weeks from Visit 2 (Day 0) to Visit 4 (Day 14) or the Early Discontinuation Visit (EDV).
Period: Overall Study
Arm/Group | Placebo | Levocetirizine
Started | 59 | 114
Safety Population | 59 | 114
Completed | 58 | 111
Not Completed | 1 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Loss of efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Levocetirizine | Total
Number analyzed (Participants) | 59 | 114 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 114 | 173
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.75 (1.45) | 3.78 (1.38) | 3.77 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 49 | 72
  Male | 36 | 65 | 101
Region of Enrollment [Number; unit: participants]
  United States | 59 | 114 | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Ventricular Rate (VR)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
beats per minute | -1.5 (14.1) | 1.3 (14.2)

2. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in RR Interval
Description: The RR interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
milliseconds | 9.2 (85.9) | -6.9 (83.4)

3. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in PR Interval
Description: The PR interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
milliseconds | 0.5 (9.6) | -0.8 (11.0)

4. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QRS Duration
Description: The QRS duration refers to the respective time duration in the Electrocardiogram (ECG).
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
milliseconds | 0.3 (6.6) | 0.9 (7.1)

5. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QT Interval
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
milliseconds | -2.8 (17.2) | -1.5 (19.2)

6. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 56 | 110
milliseconds | -5.5 (14.3) | -0.3 (16.6)

7. Primary Outcome: Absolute Value of QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) at Visit 3 (Day 7)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: 7 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 57 | 112
milliseconds | 372.6 (16.5) | 368.9 (19.4)

8. Primary Outcome: Absolute Value of QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG).
Time Frame: 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 57 | 111
milliseconds | 369.8 (17.1) | 370.5 (18.5)

9. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Total Bilirubin
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: micromole per liter [µmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 54 | 104
micromole per liter [µmol/L] | 0.000 [-10.26 to 3.42] | 0.000 [-8.55 to 5.13]

10. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Alanine Aminotransferase (ALT)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: unit per liter [U/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 54 | 105
unit per liter [U/L] | -1.5 [-12 to 167] | 1.0 [-21 to 138]

11. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Aspartate Aminotransferase (AST)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: unit per liter [U/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 53 | 105
unit per liter [U/L] | -1.0 [-15 to 52] | 1.0 [-16 to 58]

12. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Blood Urea Nitrogen
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: millimole per liter [mmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 54 | 105
millimole per liter [mmol/L] | -0.1785 [-2.142 to 2.142] | 0.0000 [-3.570 to 3.213]

13. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Blood Creatinine
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: micromole per liter [µmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 54 | 105
micromole per liter [µmol/L] | -0.8840 [-17.680 to 13.260] | 1.7680 [-15.912 to 16.796]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 1 (Day -2 to -28) over randomization and On-treatment Period up to the Follow-up Visit (Day 21±2).
Description: Adverse Events refer to the safety population including all subjects who were dispensed study treatment at least once.
Arm/Group | Placebo | Levocetirizine
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/114
Other Adverse Events (participants affected / at risk) | 21/59 | 39/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | Levocetirizine (N=114)
Pyrexia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | Levocetirizine (N=114)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Teething (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 3 (3) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.